CLINICAL TRIAL: NCT00412854
Title: Phase IIIb, Multicentre Study to Assess Safety & Immunogenicity of GSK Biologicals' Combined DTPa/Hib (Infanrix/Hib) Vaccine vs Separate Administration of DTPa (Infanrix) & Hib (Hiberix) Vaccines in Healthy Infants 3,4,&5 Months of Age as Compared With the Separate Administration of DTPa and Hib Vaccines at Different Injection Sites.
Brief Title: Study to Assess Safety & Immunogenicity of GSK Biologicals' DTPa/Hib Vaccine vs Separate Administration of DTPa and Hib.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104567
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2016-12

CONDITIONS: Tetanus; Diphtheria; Acellular Pertussis
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; Hiberix

INTERVENTIONS:
Biological: Infanrix™/Hib
Biological: Infanrix
Biological: Hiberix

SUMMARY:
This study will compare GSK Biologicals' DTPa/Hib vaccine to separately administered DTPa and Hib vaccines in Chinese infants 3, 4 & 5 months of age, in terms of safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* A male or female between, and including, 90 and 120 days of age at the time of the first vaccination,
* written informed consent obtained from the parent or guardian of the subject

Exclusion Criteria:

* Subjects with known exposure to diphtheria, tetanus, pertussis and/or Haemophilus influenzae disease can not participate,
* Subjects who have received previous vaccination against diphtheria, tetanus, acellular pertussis and/or Haemophilus influenzae type b diseases can not participate.

Ages: 90 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2007-01-03; Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- China (2):
  - GSK Investigational Site, Mengshan
  - GSK Investigational Site, Wuzhou

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Yan-Ping Li, Shumin Zhang, Qiang Ye, Qiming Hou, Yanan Li, Hong Li, Yinghua Xu, Xiao Ma, Youping Liu, Xiaoling Chen, Lirong Huang, Gunasekaran Ramakrishnan, Richard Zhao, Haiwen Tang, Olivier Van Der Meeren, Hans L Bock.Combined diphtheria-tetanus-acellular pertussis vaccine mixed with Haemophilus influenzae type b conjugate vaccine is safe and immunogenic in two studies in Chinese infants.Chinese Journal of Vaccines - Zhongguo Yi Miao He Mian Yi (Zhongguo Ji Hua Mian Yi). Zhongguo Yi Miao He Mian Yi. 2010 Apr;16(2):97-104
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104567 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Infanrix/Hib Group: Healthy male and female infants who received Infanrix/Hib vaccine as a three-dose primary vaccination course at 3, 4 and 5 months of age, administered as an intramuscular injection, into the left anterolateral thigh.
- Infanrix+Hiberix Group: Healthy male and female infants who received Infanrix and Hiberix vaccines as a three-dose primary vaccination course at 3, 4 and 5 months of age, co-administered as separate intramuscular injections, into the left and right anterolateral thighs, respectively.
Period: Overall Study
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Started | 330 | 330
Completed | 316 | 314
Not Completed | 14 | 16
Not completed — Withdrawn due to adverse events | 1 | 5
Not completed — Withdrawn for other reasons | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group | Total
Number analyzed (Participants) | 330 | 330 | 660
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 14.2 (1.12) | 14.2 (1.18) | 14.2 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 167 | 316
  Male | 181 | 163 | 344

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphteria Toxoid (D) and Tetanus Toxoid (T)
Description: A seroprotected subject was defined as a vaccinated subject with anti-D and anti-T antibody concentrations higher than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: At Month 3
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 163 | 164
Subjects
  Anti-D | 162 | 164
  Anti-T | 163 | 164
Statistical Analysis 1: Comparison: Infanrix/Hib Group vs Infanrix+Hiberix Group; Difference in seroprotection rates against diphteria toxoid: To demonstrate that the immunogenicity of Infanrix™/Hib vaccine administered at 3, 4 and 5 months of age (Infanrix/Hib Group) was non-inferior to that of the concomitant administration of Infanrix™ and Hiberix™ vaccines at the same age (Infanrix+Hiberix Group), in terms of immune response to all vaccine antigens, one month after the three-dose primary vaccination course; Test type: Non-Inferiority or Equivalence — The upper limit of the standardized asymptotic 95% confidence interval (CI) on the group difference [Infanrix+Hiberix Group minus Infanrix/Hib Group] in percentage of seroprotected subjects was ≤ 10%; Difference in seroprotection rate = 0.61, 95% CI 2-sided [-1.68 to 3.39]
Statistical Analysis 2: Comparison: Infanrix/Hib Group vs Infanrix+Hiberix Group; Difference in seroprotection rates against tetanus toxoid: To demonstrate that the immunogenicity of Infanrix™/Hib vaccine administered at 3, 4 and 5 months of age (Infanrix/Hib Group) was non-inferior to that of the concomitant administration of Infanrix™ and Hiberix™ vaccines at the same age (Infanrix+Hiberix Group), in terms of immune response to all vaccine antigens, one month after the three-dose vaccination course; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in seroprotection rate = 0.00, 95% CI 2-sided [-2.29 to 2.30]

2. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol Phosphate (PRP)
Description: A seroprotected subject was defined as a vaccinated subject with an anti-PRP antibody concentration higher than or equal to (≥) 0.15 microgram/milliliter (µg/mL).
Time Frame: At Month 3
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 162 | 164
Subjects | 158 | 164
Statistical Analysis 1: Comparison: Infanrix/Hib Group vs Infanrix+Hiberix Group; Difference in seroprotection rates against PRP: To demonstrate that the immunogenicity of Infanrix™/Hib vaccine administered at 3, 4 and 5 months of age (Infanrix/Hib Group) was non-inferior to that of the concomitant administration of Infanrix™ and Hiberix™ vaccines at the same age (Infanrix+Hiberix Group), in terms of immune response to all vaccine antigens, one month after the three-dose vaccination course; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in seroprotection rate = 2.47, 95% CI 2-sided [0.15 to 6.18]

3. Primary Outcome: Number of Subjects With a Vaccine Response to Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN) Antibodies
Description: The vaccine response was defined as it follows:
  * for PT and FHA, an antibody concentration higher than or equal to (≥) 20 EL.U/mL at post-vaccination;
  * for PRN, at least a 4-fold increase in antibody concentration from pre-vaccination to post-vaccination time points.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 163 | 164
Subjects
  Anti-PT | 163 | 164
  Anti-FHA | 163 | 164
  Anti-PRN | 159 | 162
Statistical Analysis 1: Comparison: Infanrix/Hib Group vs Infanrix+Hiberix Group; Difference in vaccine response rates against PT: To demonstrate that the immunogenicity of Infanrix™/Hib vaccine administered at 3, 4 and 5 months of age (Infanrix/Hib Group) was non-inferior to that of the concomitant administration of Infanrix™ and Hiberix™ vaccines at the same age (Infanrix+Hiberix Group), in terms of immune response to all vaccine antigens, one month after the three-dose vaccination course; Test type: Non-Inferiority or Equivalence — The upper limit of the standardized asymptotic 95% confidence interval (CI) on the group difference [Infanrix+Hiberix Group minus Infanrix/Hib Group] in percentage of subjects with a vaccine response was ≤ 10%; Difference in seroresponse rate = 0.00, 95% CI 2-sided [-2.29 to 2.30]
Statistical Analysis 2: Comparison: Infanrix/Hib Group vs Infanrix+Hiberix Group; Difference in vaccine response rates against FHA: To demonstrate that the immunogenicity of Infanrix™/Hib vaccine administered at 3, 4 and 5 months of age (Infanrix/Hib Group) was non-inferior to that of the concomitant administration of Infanrix™ and Hiberix™ vaccines at the same age (Infanrix+Hiberix Group), in terms of immune response to all vaccine antigens, one month after the three-dose vaccination course; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in seroresponse rate = 0.00, 95% CI 2-sided [-2.29 to 2.30]
Statistical Analysis 3: Comparison: Infanrix/Hib Group vs Infanrix+Hiberix Group; Difference in vaccine response rates against PRN: To demonstrate that the immunogenicity of Infanrix™/Hib vaccine administered at 3, 4 and 5 months of age (Infanrix/Hib Group) was non-inferior to that of the concomitant administration of Infanrix™ and Hiberix™ vaccines at the same age (Infanrix+Hiberix Group), in terms of immune response to all vaccine antigens, one month after the three-dose vaccination course; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in seroresponse rate = 1.23, 95% CI 2-sided [-2.17 to 5.07]

4. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ 1.0 µg/mL
Description: The number of subjects with anti-PRP antibody concentrations higher than or equal to (≥) 1.0 µg/mL post primary vaccination is reported.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 162 | 164
Subjects | 145 | 156

5. Secondary Outcome: Concentrations for Anti-D and Anti-T Antibodies
Description: Anti-D and anti-T antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in International units per milliliter (IU/mL).
Time Frame: At Month 0 and Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 163 | 164
IU/mL
  Anti-D (Month 0) | 0.050 [0.050 to 0.051] | 0.051 [0.050 to 0.052]
  Anti-D (Month 3) | 0.545 [0.505 to 0.588] | 0.567 [0.530 to 0.606]
  Anti-T (Month 0) | 0.050 [0.050 to 0.050] | 0.050 [0.050 to 0.051]
  Anti-T (Month 3) | 2.990 [2.858 to 3.127] | 3.214 [3.091 to 3.341]

6. Secondary Outcome: Concentrations for Anti-PRP Antibodies
Description: Anti-PRP antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in microgram/milliliter (µg/mL).
Time Frame: At Month 0 and Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 163 | 164
µg/mL
  Anti-PRP, Month 0 (N=163;164) | 0.083 [0.076 to 0.092] | 0.083 [0.078 to 0.088]
  Anti-PRP, Month 3 (N=162;164) | 3.559 [3.003 to 4.219] | 6.120 [5.355 to 6.995]

7. Secondary Outcome: Concentrations for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 163 | 164
EL.U/mL
  Anti-PT | 66.0 [61.5 to 70.8] | 67.0 [62.5 to 71.8]
  Anti-FHA | 207.2 [192.2 to 223.4] | 198.1 [182.7 to 214.8]
  Anti-PRN | 172.4 [157.9 to 188.3] | 177.5 [163.3 to 192.9]

8. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) follow-up period after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one study vaccine administration documented and with the symptoms sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 323 | 326
Subjects
  Any Pain, Dose 1 (N=323;326) | 44 | 46
  Grade 3 Pain, Dose 1 (N=323;326) | 2 | 3
  Any Redness, Dose 1 (N=323;326) | 5 | 11
  Grade 3 Redness, Dose 1 (N=323;326) | 0 | 0
  Any Swelling, Dose 1 (N=323;326) | 3 | 1
  Grade 3 Swelling, Dose 1 (N=323;326) | 1 | 0
  Any Pain, Dose 2 (N=317;313) | 23 | 32
  Grade 3 Pain, Dose 2 (N=317;313) | 0 | 0
  Any Redness, Dose 2 (N=317;313) | 3 | 11
  Grade 3 Redness, Dose 2 (N=317;313) | 2 | 0
  Any Swelling, Dose 2 (N=317;313) | 9 | 7
  Grade 3 Swelling, Dose 2 (N=317;313) | 1 | 0
  Any Pain, Dose 3 (N=316;312) | 19 | 25
  Grade 3 Pain, Dose 3 (N=316;312) | 1 | 0
  Any Redness, Dose 3 (N=316;312) | 7 | 8
  Grade 3 Redness, Dose 3 (N=316;312) | 1 | 0
  Any Swelling, Dose 3 (N=316;312) | 8 | 6
  Grade 3 Swelling, Dose 3 (N=316;312) | 2 | 0
  Any Pain, Across doses (N=323;326) | 59 | 71
  Grade 3 Pain, Across doses (N=323;326) | 3 | 3
  Any Redness, Across doses (N=323;326) | 14 | 24
  Grade 3 Redness, Across doses (N=323;326) | 2 | 0
  Any Swelling, Across doses (N=323;326) | 17 | 13
  Grade 3 Swelling, Across doses (N=323;326) | 4 | 0

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.1 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever above (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after each vaccine dose and across doses
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 323 | 327
Subjects
  Any Drowsiness, Dose 1 (N=323;327) | 71 | 84
  Grade 3 Drowsiness, Dose 1 (N=323;327) | 0 | 3
  Related Drowsiness, Dose 1 (N=323;327) | 59 | 72
  Any Fever (Axillary), Dose 1 (N=323;327) | 105 | 141
  Grade 3 Fever (Axillary), Dose 1 (N=323;327) | 0 | 0
  Related Fever (Axillary), Dose 1 (N=323;327) | 93 | 130
  Any Irritability, Dose 1 (N=323;327) | 125 | 123
  Grade 3 Irritability, Dose 1 (N=323;327) | 1 | 2
  Related Irritability, Dose 1 (N=323;327) | 111 | 107
  Any Loss of appetite, Dose 1 (N=323;327) | 69 | 79
  Grade 3 Loss of appetite, Dose 1 (N=323;327) | 0 | 2
  Related Loss of appetite, Dose 1 (N=323;327) | 53 | 63
  Any Drowsiness, Dose 2 (N=317;313) | 49 | 45
  Grade 3 Drowsiness, Dose 2 (N=317;313) | 0 | 1
  Related Drowsiness, Dose 2 (N=317;313) | 45 | 42
  Any Fever (Axillary), Dose 2 (N=317;313) | 82 | 106
  Grade 3 Fever (Axillary), Dose 2 (N=317;313) | 0 | 0
  Related Fever (Axillary), Dose 2 (N=317;313) | 79 | 104
  Any Irritability, Dose 2 (N=317;313) | 78 | 84
  Grade 3 Irritability, Dose 2 (N=317;313) | 1 | 3
  Related Irritability, Dose 2 (N=317;313) | 74 | 82
  Any Loss of appetite, Dose 2 (N=317;313) | 55 | 51
  Grade 3 Loss of appetite, Dose 2 (N=317;313) | 0 | 0
  Related Loss of appetite, Dose 2 (N=317;313) | 48 | 47
  Any Drowsiness, Dose 3 (N=316;312) | 29 | 25
  Grade 3 Drowsiness, Dose 3 (N=316;312) | 0 | 1
  Related Drowsiness, Dose 3 (N=316;312) | 26 | 22
  Any Fever (Axillary), Dose 3 (N=316;312) | 81 | 91
  Grade 3 Fever (Axillary), Dose 3 (N=316;312) | 1 | 0
  Related Fever (Axillary), Dose 3 (N=316;312) | 72 | 84
  Any Irritability, Dose 3 (N=316;312) | 55 | 67
  Grade 3 Irritability, Dose 3 (N=316;312) | 1 | 1
  Related Irritability, Dose 3 (N=316;312) | 51 | 60
  Any Loss of appetite, Dose 3 (N=316;312) | 45 | 41
  Grade 3 Loss of appetite, Dose 3 (N=316;312) | 0 | 0
  Related Loss of appetite, Dose 3 (N=316;312) | 39 | 38
  Any Drowsiness, Across doses (N=323;327) | 104 | 109
  Grade 3 Drowsiness, Across doses (N=323;327) | 0 | 5
  Related Drowsiness, Across doses (N=323;327) | 93 | 99
  Any Fever (Axillary), Across doses (N=323;327) | 174 | 201
  Grade 3 Fever (Axillary), Across doses (N=323;327) | 1 | 0
  Related Fever (Axillary), Across doses (N=323;327) | 164 | 193
  Any Irritability, Across doses (N=323;327) | 161 | 170
  Grade 3 Irritability, Across doses (N=323;327) | 3 | 6
  Related Irritability, Across doses (N=323;327) | 150 | 154
  Any Loss of appetite, Across doses (N=323;327) | 120 | 120
  Grade 3 Loss of appetite, Across doses (N=323;327) | 0 | 2
  Related Loss of appetite, Across doses (N=323;327) | 103 | 105

10. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-30) follow-up period after each vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least one study vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 330 | 328
Subjects | 171 | 189

11. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From receipt of first dose of study vaccine (Day 0) to study end (Month 3)
Population: as for outcome 10
Measure: Number; unit: Subjects
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Number analyzed (Participants) | 330 | 328
Subjects | 4 | 7

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Day 0-3) follow-up period; Unsolicited AEs: within 31 days (Day 0-30) post-vaccination; SAEs: during the entire study period (from Day 0 to Month 3).
Arm/Group | Infanrix/Hib Group | Infanrix+Hiberix Group
Serious Adverse Events (participants affected / at risk) | 4/330 | 7/328
Other Adverse Events (participants affected / at risk) | 278/330 | 290/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix/Hib Group (N=330) | Infanrix+Hiberix Group (N=328)
Bronchopneumonia (Infections and infestations) | 1 | 3
Bronchitis (Infections and infestations) | 2 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Hemorrhage (Vascular disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infanrix/Hib Group (N=330) | Infanrix+Hiberix Group (N=330)
Pain (General disorders) | 59/323 | 71
Redness (General disorders) | 14/323 | 24
Swelling (General disorders) | 17/323 | 13
Drowsiness (General disorders) | 104/323 | 109
Fever (Axillary) (General disorders) | 174/323 | 201
Irritability (General disorders) | 161/323 | 170
Loss of appetite (General disorders) | 120/323 | 120
Nasopharyngitis (Infections and infestations) | 119 | 127
Diarrhea (Gastrointestinal disorders) | 38 | 39
Pyrexia (General disorders) | 17 | 23

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.